CLINICAL TRIAL: NCT00641121
Title: Bethaherpesviruses in Children Who Are Immune Suppressed
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Johanna Goldfarb, Contract Staff, The Cleveland Clinic
Other Study IDs: 7689
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Immune Suppressed Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Unexplained fever in children with cancer is a common occurrence, often requiring hospital admission for evaluation and treatment with intravenous antibiotics. While empiric use of intravenous antibiotics is the norm in this population, between 48-70% of febrile and neutropenic episodes remain without an identifiable source. An understudied area is the potential role of betaherpesvirus infections in such febrile episodes. These viruses are significant pathogens in patients who become immunocompromised in conjunction with organ transplantation or acquired immune deficiency syndrome (AIDS). It is possible that they are similarly pathogenic in children who become immunocompromised due to cancer chemotherapy.

Thus, we will investigate the association between the betaherpesviruses and fever in children with cancer. The betaherpesviruses include cytomegalovirus (CMV), human herpesvirus 6A (HHV-6A), human herpesvirus 6B (HHV-6B), and human herpesvirus 7 (HHV-7). These viruses are grouped based on shared biological and genetic properties. Each is commonly acquired in childhood, persists in the human host, and can reactivate. Reactivation occurs intermittently throughout life in healthy individuals and is seldom associated with disease. Immune suppression is associated with a higher likelihood of reactivation and clinical disease. Latency of these viruses involves highly regulated processes that result in the viruses evading destruction and persisting within the host. Should balance be disrupted, as with cancer and anticancer therapy altering the normal host state, the environment may become favorable for betaherpesvirus reactivation, leading to disease and further alterations of the immune system.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with cancer (leukemia, lymphoma, or solid tumor)
2. Undergoing solid organ pre-transplantation evaluation
3. Age birth to 21 years

Exclusion Criteria:

1. Unwilling to participate in the study
2. Unwilling to have specimens stored for future research
3. Clinical conditions preclude the required amount of blood to be drawn for the study
4. Patient has malignancy that has relapsed
5. Patient is not a primary transplant candidate (ie. has already had a solid organ transplant) -

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Chilren that are Immune suppressed
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Goldfarb, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States